# National Longitudinal Cohort of Hematological Diseases - Aplastic Anemia

(NICHE-AA)

## **Statistical Analysis Plan**

Applicant: Institute of Hematology & Blood Diseases Hospital

Version: 1.0

NCT Number: NCT04645199

Date: 4-December-2020

National Longitudinal Cohort of Hematological Diseases- Aplastic Anemia (NICHE-AA)

### Statistical Analysis Plan

# National Longitudinal Cohort of Hematological Diseases - Hemophilia

(NICHE- Hemophilia)

**Statistical Analysis Plan** 

Applicant: Institute of Hematology & Blood Diseases Hospital

Version: 1.0

NCT Number: NCT04645199

Date: 27-August-2020

National Longitudinal Cohort of Hematological Diseases- Hemophilia (NICHE-Hemophilia)

### Statistical Analysis Plan

# National Longitudinal Cohort of Hematological Diseases - Acute Myeloid Leukemia (NICHE- AML)

**Statistical Analysis Plan** 

Applicant: Institute of Hematology & Blood Diseases Hospital

Version: 1.0

NCT Number: NCT04645199

Date: 30-July-2020

National Longitudinal Cohort of Hematological Diseases-Acute Myeloid Leukemia (NICHE-AML)

#### **Statistical Analysis Plan**

# National Longitudinal Cohort of Hematological Diseases - Multiple Myeloma (NICHE- MM)

## **Statistical Analysis Plan**

Applicant: Institute of Hematology & Blood Diseases Hospital

Version: 1.0

NCT Number: NCT04645199

Date: 30-July-2020

National Longitudinal Cohort of Hematological Diseases- Multiple Myeloma (NICHE-MM)

### Statistical Analysis Plan